CLINICAL TRIAL: NCT06374771
Title: Analgesic Effect of Melatonin and Vitamin C Administration, Alone or In Combination in Major Abdominal Surgery. A Randomized Double-blind Study
Brief Title: Analgesic Effect of Melatonin and Vitamin C Administration, Alone or In Combination in Major Abdominal Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Amr Kamal Zahran, Associate Professor of Anesthesia, intensive care medicine and Pain therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-15-2022
Record Dates: First submitted 2024-04-14; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Melatonin; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Melatonin (M group) (Active Comparator): Two hours before surgery, patients will receive 10 mg of melatonin (Melatonin 10 mg - Puritan's Pride premium company) orally which will be continued once daily for 3 days postoperative at the same time as the first administration.
  Interventions: Drug: Melatonin 10 MG
- Vitamin C (V group) (Active Comparator): Two hours before surgery, patients will receive 1gm of vitamin C (Sanso C 1000 mg - AUG pharma company) orally which will be continued once daily for 3 days postoperative at the same time as the first administration.
  Interventions: Drug: Vitamin C
- Melatonin and Vitamin C (VM group) (Active Comparator): Two hours before surgery, patients will receive 10mg of melatonin and 1gm of vitamin C orally which will be continued once daily for 3 days postoperative at the same time as the first administration.
  Interventions: Drug: Melatonin 10 MG; Drug: Vitamin C

INTERVENTIONS:
Drug: Melatonin 10 MG — 10 mg of Melatonin will be given orally pre and post-operative
  Other Names: (Melatonin 10 mg - Puritan's Pride premium company)
  Arms: Melatonin (M group); Melatonin and Vitamin C (VM group)
Drug: Vitamin C — 1 gm of Vitamin C will be given orally pre and post-operative
  Other Names: (Sanso C 1000 mg - AUG pharma company)
  Arms: Melatonin and Vitamin C (VM group); Vitamin C (V group)

SUMMARY:
The goal of this clinical trial is to compare the analgesic effect of melatonin, and vitamin C and their combination in patients aged 18-60 years old who will undergo major abdominal surgery with mid-line incision within an expected time of surgery from 3 to 5 hours e.g. radical cystectomy, radical prostatectomy, colectomy, sigmoidectomy, splenectomy, and CBD exploration through mid-line incision.

This study hypothesizes that using both vitamin C and melatonin together as adjuvants will cause:

* More reduction in total morphine consumption in the first 24 hours postoperatively
* More reduction of the incidence of chronic post-surgical pain, than using each adjuvant alone.

Participants will be allocated into three equal groups: Melatonin (M group) and vitamin C (V group), and Melatonin and vitamin C (VM group). Two hours before surgery all patients will receive the study drugs orally and will be continued for 3 days postoperative at the same time of the first administration; 10mg of melatonin for M group (Melatonin 10 mg - Puritan's Pride premium company), 1gm of vitamin C for V group (Sanso C 1000 mg - AUG pharma company), and 10mg of melatonin and 1gm of vitamin C for VM group.

Researchers will compare:

* The effect of melatonin, vitamin C, and their combination on postoperative opioid consumption
* The severity of postoperative pain, using the Numerical Rating Scale (NRS)
* Patients' satisfaction with a three-point scale
* The time of the first requirement for rescue analgesia
* The effect on the incidence of chronic post-surgical pain.

DETAILED DESCRIPTION:
Randomization will be performed using computer-generated numbers with Random Allocation Software (https://random-allocation-software.software.informer.com/2.0/), in a 1:1:1 ratio. 60 consequentially numbered opaque envelopes (20 per group) will be made containing group assignments and drug administration instructions. A research assistant will be responsible for opening the envelopes and the assigned drug administration without further involvement in the study. A blinded anesthesiologist will be responsible for the anesthetic management, perioperative data collection, and postoperative pain assessment and analgesia administration.

A full history will be taken from all patients. Age, sex, height, weight, and the American Society of Anesthesiologists' (ASA) score will be recorded.

Preoperatively, patients' laboratory investigations as complete blood count, prothrombin time, concentration and INR, liver function tests, and kidney function tests will be recorded. Clinical assessment will be carried out for their eligibility for the study.

Patients will be allocated into three equal groups: Melatonin (M group) and vitamin C (V group), and Melatonin and vitamin C (VM group). Two hours before surgery all patients will receive the study drugs orally and will be continued for 3 days postoperative at the same time of the first administration [10], 10mg of melatonin for M group (Melatonin 10 mg - Puritan's Pride premium company), 1gm of vitamin C for V group (Sanso C 1000 mg - AUG pharma company), and 10mg of melatonin and 1gm of vitamin C for VM group.

The patients will attend the pre-anesthesia room one hour before the procedure, NRS pain score (Figure 1) will be explained to all candidates (zero corresponds to no pain and 10 is indicative of the worst unbearable pain).

Baseline vital signs will be then recorded including non-invasive measurements of systolic, mean, diastolic arterial blood pressures, heart rate, and oxygen saturation.

Anesthetic technique Upon arrival at the operating room, standard monitoring (non-invasive blood pressure, electrocardiography, and pulse oximetry) will be applied. The patient will receive pre-induction ondansetron 8mg as an antiemetic drug. Anesthesia will be induced using propofol 1-2 mg/kg, fentanyl 2 µg/kg, and lidocaine 1 mg/kg. Atracurium 0.5 mg/kg will be administered to facilitate endotracheal intubation. After intubation, the capnography will be connected and the patients will be mechanically ventilated to maintain end-tidal CO2 between 30-35 mmHg. Anesthesia will be maintained with sevoflurane inhalational anesthetic in 50% oxygen and top-up doses of atracurium 0.1mg/kg every 20 minutes to maintain muscle relaxation. After the skin incision, a bolus dose of morphine100mcg/kg will be given. Fentanyl at 1µg/kg will be administered as rescue analgesia if an intraoperative increase in heart rate or systolic blood pressure by 20% occurs, after the exclusion of other causes rather than pain. Before skin closure, paracetamol 1gm will be given intravenously. Depth of anesthesia will be monitored by a bispectral index monitoring device (BIS) to maintain the readings within 40 to 55, all through the procedure. Mean blood pressure and heart rate are maintained within ±20%.

Postoperative Technique:

Pain will be classified as mild (NRS 0-4), moderate (NRS 5-7), and severe (NRS 8-10). Recovery time is defined as the time from extubation to the time of achieving Aldrete scores ≥ 9. The patient is transferred to the post-anesthesia care unit (PACU); Blood pressure, heart rate, and oxygen saturation will be monitored every 15 minutes till discharge from the PACU. In PACU, a bolus dose of morphine; the physician will give 50 mcg/kg if the pain score of the patient is > 4. All patients with a numeric score ≤ 4 will receive morphine via an infusion pump (Zhejiang Fert disposable infusion pump 275ml with constant flow 5ml/hour. Zhejiang Fert Medical Device Co., Ltd). They will receive a morphine continuous infusion of 10mcg/kg/hour (maximum 1 mg/hour). The patients will be instructed to report any pain to a pain nurse, and if the NRS increases to more than 4, the pain nurse will inform the anesthesiologist. Inadequate analgesia (NRS >4) will be treated with a clinician bolus of 50mcg/kg with a time interval of 30 minutes at least between the additional doses till NRS decreases to less than 4. Excessive somnolence or respiratory depression will be treated by stopping the pump until appropriate recovery and by a decrease in the demand dose of 20%. Paracetamol 1gm will be administered every 8 hours intravenously.

Postoperative, hemodynamics including systolic and diastolic blood pressures (SBP and DBP), heart rate (HR), SpO2, NRS, Richmond Agitation Sedation Scale (RASS) and patient satisfaction (using Likert three-point scale; good, moderate, and bad) scores will be recorded at 2, 4, 6, 12, 24 hours. The total morphine consumption including the continuous infusion, total boluses required, and the number of boluses will be recorded at the end of the first 24 hours.

The side effects of opioids will be recorded; e.g. nausea, vomiting, pruritus, urine retention, and allergic reactions. In case of vomiting, metoclopramide 10 mg will be given. Ondansetron 8mg will be given in persistent vomiting. In the case of respiratory depression, Naloxone 1mcg/kg will be administered and oxygen will be supplied through an oxygen mask.

NRS and patient satisfaction using a Likert 3-point scale will be recorded from the patient after 48, 72, 96 h, one month, and 3 months post-operative.

Three months follow-up phase assessment parameters:

Chronic pain assessments will be conducted during patients' visits to the pain clinic in the first and third postoperative months by a blinded physician and include the following:

1. the location, intensity, nature, and duration of pain as well as any aggravating or mitigating factors,
2. Analgesic medication used
3. For cancer patients, adjuvant treatment used (e.g., chemotherapy and radiotherapy) Chronic Neuropathic pain will be assessed using the Numeric Pain Rating Scale

Data collection:

* All hemodynamic parameters such as blood pressure using non-invasive measurement, heart rate, and oxygen saturation will be recorded every 10 minutes from skin incision to skin closure and at 2, 4 h postoperatively. Other complications such as hypotension, nausea, and vomiting will be monitored and recorded.
* Postoperative morphine consumption during the first 24 hours.
* NRS pain score immediately postoperatively and then at 30 minutes, 2, 4, 6, 12,24, 48, 72, 96 hours one month and three months. NRS will also be recorded when the patient begins to move. Dynamic pain will be defined as the difference in NRS score between rest and walking >2 points. Pain will be classified as mild (NRS 0-4), moderate (NRS 5-7), and severe (NRS 8-10).
* RASS score immediately postoperatively and then at 30 minutes, 2, 4, 6, 12, and 24 hours.
* Patient's satisfaction Likert three-point scale on the first postoperative day,48, 73, 96 hours, one month, and three months.
* Postoperative opioid-related complications (e.g. Nausea, vomiting, constipation, sedation).
* Anesthesia time starting from induction of anesthesia till extubation of the patient.
* Surgical operation time starting from skin incision till skin closure.
* Emergence time is defined as from discontinuation of inhalational anesthesia till the extubation of the patient
* Recovery time is defined as the time from extubation to the time of achieving Aldrete scores ≥ 9

ELIGIBILITY:
Inclusion Criteria:

* ASA I -II
* Expected time of operation 3-5 hours

Exclusion Criteria:

* BMI > 35 kg/m2
* Presence of psychiatric or mental disorders.
* Chronic pain syndromes (neuropathic pain, post-herpetic neuralgia, Complex regional pain syndrome)
* Drug or alcohol abuse.
* Hepatic failure (Child class B- Child class C)
* Renal impairment (creatinine > 2mg/dL or CKD on regular dialysis)
* History of any allergic reaction to the drugs used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-27 (Estimated); Primary Completion 2024-06-27 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | The 1st 24 postoperative hours
  mg

SECONDARY OUTCOMES:
Numeric Rating Scale | 5 minutes after extubation, 30 minutes, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, one month and three months
  Pain will be classified as mild (NRS 0-4), moderate (NRS 5-7), and severe (NRS 8-10)
Richmond Agitation Sedation Scale | 5 minutes after extubation, 30 minutes, 2 hours, 4 hours, 6 hours, 12 hours and 24 hours
  (-5) Unarousable, (-4) Deep sedation, (-3) Moderate sedation, (-2) Light sedation, (-1) Drowsy, (0) Alert and calm, (+1) Restless, (+2) Agitated, (+3) Very agitation, and (+4) Combative
Time to first analgesic request | from the time of end of surgery till the first analgesic requirement during the 24 hours postoperative
  minutes
chronic post-surgical pain | 3 months
  present or not present
patient satisfaction using Likert three-point scale | 24 hours, 48 hours, 72 hours, 96 hours, one month and three months postoperative
  good, moderate, or bad
systolic blood pressure | every 10 minutes from skin incision to skin closure and at 2, 4 hours post operatively.
  mmHg
Heart rate | every 10 minutes from skin incision to skin closure and at 2, 4 hours post operatively.
  beat per minute
Intra-operative mean consumption of sevoflurane per hour. | from the start of anesthesia till the end of anesthesia
  ml per hour

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Hamimy, MD, Study Chair — Professor of Anesthesiology
Locations (1):
- Faculty of Medicine - Cairo University, Cairo, Manial, Egypt